CLINICAL TRIAL: NCT00491725
Title: A Multi-centre, Single Armed, Open Labelled Trial to Study the Efficacy and Safety Profile of Repaglinide & Metformin Combination Therapy in Chinese Type 2 Diabetics
Brief Title: Efficacy and Safety of Repaglinide and Metformin Combination Therapy in Type 2 Diabetes Failing on Oral Anti-diabetic Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1655
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repaglinide
Drug: metformin

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate the efficacy and safety of repaglinide and metformin combination therapy in Chinese subjects with type 2 diabetes inadequately controlled with OAD (oral anti-diabetic drugs).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 weeks
* HbA1c: 8.0-10.0%
* Current treatment with OAD on monotheray or OAD on combination therapy
* Body mass index (BMI): 21.0-35.0 kg/m2

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Recurrent major hypoglycaemia as judged by the Investigator
* Uncontrolled hypertension
* Any other significant condition or concomitant disease such as endocrine, cardiac, neurological, malignant or other pancreatic disease as judged by the Investigator

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 18 weeks of treatment

SECONDARY OUTCOMES:
Post Prandial Plasma Glucose
Fasting Plasma Glucose (FPG)
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com